CLINICAL TRIAL: NCT05934942
Title: An Open-label, Fixed-sequence Cross-over, Two-period, Phase I Trial to Evaluate the Effect of Multiple Doses of BI 1358894 on the Pharmacokinetics of a Combination of Ethinylestradiol and Drospirenone in Healthy Female Subjects
Brief Title: A Study in Healthy Women to Test Whether BI 1358894 Influences the Amount of a Contraceptive in the Blood
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1402-0019
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination; TRPC inhibitor BI 1358894

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yasmin® (Reference treatment (R)) followed by BI 1358894 and Yasmin® (Test treatment (T)) (Experimental): All female participants were treated with 1 daily tablet of the contraceptive Yasmin® (ethinylestradiol and drospirenone) during the run-in period (Day-56 to Day-8).
  Since the study was discontinued as per protocol after the run-in period, none of the participants received the intended treatments for periods 1 and 2.
  Interventions: Drug: Yasmin®; Drug: BI 1358894

INTERVENTIONS:
Drug: Yasmin® — Ethinylestradiol (EE) and Drospirenone (DRSP)
Drug: BI 1358894 — BI 1358894

SUMMARY:
This study aims to investigate the effect of multiple doses of BI 1358894 on pharmacokinetics of ethinylestradiol (EE) and drospirenone (DRSP) (Yasmin®)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy premenopausal female subjects according to the assessment of the investigator, as based on a complete medical history including a physical and gynaecological examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 35 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
5. Female subject who meet any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

   * Use of an oral hormonal contraception method in combination with a barrier contraception method and willing to stop the hormonal method and to continue using the barrier method plus Yasmin® for the duration of the trial
   * Use of non-hormonal intrauterine device (IUD)
   * Sexually abstinent
   * Female subject who underwent tubal ligation
   * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator (e.g. pronounced varicosis, thrombophlebitis, and evidence of peripheral circulatory disturbances)
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts

Further exclusion criteria apply

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomized, open-label, two-period, fixed-sequence trial involving a run-in phase. The study treated 28 healthy female participants with Yasmin® in the run-in period and aimed to compare Yasmin® (reference treatment) with the combination of Yasmin® and BI 1358894 (test treatment).
Pre-assignment Details: 29 female participants of child-bearing potential who met all inclusion and no exclusion criteria entered the study, 28 were treated with Yasmin® , 1 was not treated, and 1 withdrew. 27 participants completed the run-in period. No female participant received an investigational medicinal treatment in Period 1 (Yasmin® alone) or Period 2 (Yasmin® and BI 1358894). The study was prematurely discontinued as per protocol in the run-in period.
Groups:
- Yasmin® (Reference Treatment) Followed by BI 1358894 and Yasmin® (Test Treatment): All female participants were treated with 1 daily tablet of the contraceptive Yasmin® (ethinylestradiol and drospirenone) during the run-in period (Day-56 to Day-8).
  The study was discontinued as per protocol in the run-in period, and thus none of the participants received the planned treatments for period 1 (reference treatment (R)) and for period 2 (test treatment (T)).
  Period 1: The planned reference treatment was to administer one tablet of Yasmin® daily after a continental breakfast on Days 1-21 of period 1 (not administered).
  Period 2: The planned test treatment consisted of one tablet of Yasmin®, one tablet of BI 1358894 25 milligram (mg) and two tablets of BI 1358894 50 mg (for a total dose of BI 1358894 = 125mg) each administered daily after a continental breakfast on Days 1-21 in period 2 (not administered).
Period: Run-in Period
Arm/Group | Yasmin® (Reference Treatment) Followed by BI 1358894 and Yasmin® (Test Treatment)
Started | 29
Completed | 27
Not Completed | 2
Not completed — Not treated | 1
Not completed — Withdrawal by Subject | 1
Period: Period 1 - Reference Treatment
Arm/Group | Yasmin® (Reference Treatment) Followed by BI 1358894 and Yasmin® (Test Treatment)
Started | 0 (The study was discontinued as per protocol after the run-in period, none of the participants received the planned treatments for period 1 and 2.)
Completed | 0
Not Completed | 0
Period: Period 2 - Test Treatment
Arm/Group | Yasmin® (Reference Treatment) Followed by BI 1358894 and Yasmin® (Test Treatment)
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All subjects who were entered to the trial and received Yasmin® during the run-in period.
Arm/Group | Yasmin® (Reference Treatment) Followed by BI 1358894 and Yasmin® (Test Treatment)
Number analyzed (Participants) | 28
Age, Customized [Median (Full Range); unit: Years] | 30 [22 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Ethinylestradiol and Drospirenone in Plasma at Steady State Over the Uniform Dosing Interval τ (AUCτ,ss)
Time Frame: Planned: pre-dose within 10 minutes before 1st drug administration, and then in period 1 and period 2 post-dose : 480:30, 481:00, 481:30, 482:00, 482:30, 483:00, 483:30, 484:00, 485:00, 486:00, 488:00, 490:00, 492:00, 504:00 hours (h)
Population: The study was prematurely discontinued as per protocol after run-in period. No pharmacokinetic (PK) parameter values were collected. Therefore, the PK parameter analysis set as defined in the protocol was not applicable.
Groups:
- Yasmin® (Reference Treatment): All female participants were treated with 1 daily tablet of the contraceptive Yasmin® (ethinylestradiol and drospirenone) during the run-in period (Day-56 to Day-8).
  The study was discontinued as per protocol in the run-in period, and thus none of the participants received the planned treatments for period 1 (reference treatment (R)) and for period 2 (test treatment (T)).
  Period 1: The planned reference treatment was to administer one tablet of Yasmin® daily after a continental breakfast on Days 1-21 of period 1 (not administered).
- BI 1358894 and Yasmin® (Test Treatment): All female participants were treated with 1 daily tablet of the contraceptive Yasmin® (ethinylestradiol and drospirenone) during the run-in period (Day-56 to Day-8).
  The study was discontinued as per protocol in the run-in period, and thus none of the participants received the planned treatments for period 1 (reference treatment (R)) and for period 2 (test treatment (T)).
  Period 2: The planned test treatment consisted of one tablet of Yasmin®, one tablet of BI 1358894 25 milligram (mg) and two tablets of BI 1358894 50 mg (for a total dose of BI 1358894 = 125mg) each administered daily after a continental breakfast on Days 1-21 in period 2 (not administered).
Arm/Group | Yasmin® (Reference Treatment) | BI 1358894 and Yasmin® (Test Treatment)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Maximum Measured Concentration of Ethinylestradiol and Drospirenone in Plasma at Steady State Over the Uniform Dosing Interval τ (Cmax,ss)
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Yasmin® (Reference Treatment) | BI 1358894 and Yasmin® (Test Treatment)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Minimum Measured Concentration of Ethinylestradiol and Drospirenone in Plasma at Steady State Over the Uniform Dosing Interval τ (Cmin,ss)
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Yasmin® (Reference Treatment) | BI 1358894 and Yasmin® (Test Treatment)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Run-in period (Yasmin® only): Adverse events and all-cause mortality: From first Yasmin® administration on Day -56 until last administration of Yasmin® on Day -8 plus 9 days (residual effect period), up to 57 days.
Description: Treated set: All subjects who were entered to the trial and received Yasmin® during the run-in period.
Groups:
- Yasmin® (run-in Period): All female participants were treated with 1 daily tablet of the contraceptive Yasmin® (ethinylestradiol and drospirenone) during the run-in period (Day-56 to Day-8).
  Since the study was discontinued as per protocol in the run-in period, none of the participants received the intended treatments for periods 1 and 2.
Arm/Group | Yasmin® (run-in Period)
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 9/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Yasmin® (run-in Period) (N=28)
Nasopharyngitis (Infections and infestations) | 3
Headache (Nervous system disorders) | 4
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued as per protocol during the run-in period and no data for the primary and secondary pharmacokinetic endpoints could be collected, and the statistical evaluations were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT05934942/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT05934942/SAP_001.pdf